CLINICAL TRIAL: NCT05825677
Title: Investigating Stress-Induced Dopamine Release: a fMRI-PET Study
Acronym: ISIDORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2022-A00907-36
Record Dates: First submitted 2023-03-28; First posted 2023-04-24 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Stress Response
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Intervention Model Description: In a randomized controlled double-blind study, 30 healthy subjects, will be randomly assigned to 2 groups. A group of 15 participants will receive 30 minutes of active tDCS (1mA, 30 minutes with the anode at the left DLPFC and the cathode at the right DLPFC); a group of 15 participants will receive 30 minutes of placebo stimulation. All participant will be in a PET-MRI scanner for 110min, during which they will undergo the stimulation (either active or sham). During this stimulation session, all participants will undergo a standardized stress test combining psychosocial stress and physical stress.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subject will be blind of the treatment he receives (active or placebo). The experimenter, caregiver and investigator will also be blinded from stimulation (active or placebo).
  Each subject will be assigned a randomization code, corresponding to the code to enter the tDCS device. This system allows the person who administers tDCS and the subject receiving the stimulation to be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Active brain stimulation Direct current stimulation of DLPFC for 30min with an intensity of 1mA
  Interventions: Device: tDCS actif
- Sham tDCS (Sham Comparator): Sham brain stimulation Direct current stimulation of DLPFC for 30sec with an intensity of 1mA
  Interventions: Device: tDCS Sham

INTERVENTIONS:
Device: tDCS actif — Active brain stimulation
  Arms: Active tDCS
Device: tDCS Sham — Sham brain stimulation
  Arms: Sham tDCS

SUMMARY:
The stress response is mediated by the activation of the hypothalamo-pituitary-adrenal axis and the sympathetic nervous system, leading to glucocorticoid and catecholamines release respectively. This stress response is regulated by feedback loops, involving cortical and subcortical structures.

Non-invasive brain stimulation applied over the dorsolateral prefrontal cortex modulates the subcortical dopaminergic transmission at rest and can reduce the hormonal and cognitive alterations induced by stress. This study aims to investigate the Non-invasive brain stimulation -induced modulation of dopamine transmission in an acute stress situation.

DETAILED DESCRIPTION:
Objective: to investigate the influence of Dorsolateral Prefrontal Cortex stimulation during acute stress on the subcortical dopamine transmission in healthy subjects.

Method: 30 healthy subjects will be enrolled and randomized into 2 parallel groups. 15 participants will receive active Transcranial direct current stimulation , the other 15 participants will receive sham Transcranial direct current stimulation.

Transcranial direct current stimulation procedure: active Transcranial direct current stimulation corresponds to 30min of stimulation at 1mA intensity . The sham stimulation corresponds to 30s of real stimulation.

Stress paradigm: In order to induce moderate stress in humans in laboratory condition, the investigators will use the Maastricht Acute Stress test . This test is a combination between physical, hand immersion in cold water and cognitive calculation stress. The test will start 5 minutes after the beginning of stimulation session.

Stress measures: the stress response will be evaluated at the following levels:

* Neurochemical level: dopamine transmission measured with positron emission tomography
* Functional brain connectivity: resting-state networks measured with functional magnetic resonance imaging
* Hormonal level: adrenocorticotropic hormone and cortisol levels measured with blood samples
* Cognitive level: decision-making and memory assessed with delay-discounting task and reality-monitoring task, respectively
* Molecular level: expression of genes involved in the glucocorticoid receptor signaling pathway measured through blood samples Exploratory measure: Brain-Derived Neurotrophic Factor and cytoplasmic catechol-O-methyltransferase polymorphisms of participants involved in differential Transcranial direct current stimulation response will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* - Men and women aged between 18- and 30-year-old
* Non-smoker
* Non-psychotropic user

Exclusion Criteria:

* - Have a psychiatric or somatic disorder
* Have a first-degree family history of a psychiatric disorder
* Pregnant or nursing women
* Be on medication, with the exception of oral contraceptives
* Contraindications to tDCS or MRI examination
* Participants with pacemaker or cardiac or cerebral implant

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Dopamine transmission measured with positron emission tomography | One year
  Subcortical dopaminergic transmission will be analyzed, using [11C]raclopride PET activity (D2 receptor antagonist)

SECONDARY OUTCOMES:
Functional brain connectivity | One year
  Resting-state functional connectivity
Hormonal stress reactivity | One year
  ACTH level will be measured
Cognitive stress reactivity | One year
  Decision-making capacities will be measured using a computerized version of the DDT in which participants have to choose between 2 rewards. Memory capacities will be measured using a computerized task evaluating reality-memory.
Expression of genes involved in the glucocorticoid receptor signaling pathway measured through blood samples | One year
  Expression rates of genes involved in the glucocorticoid receptor signaling pathway
Assessment of brain-derived neurotrophic factor before and after transcranial direct current stimulation. | One year
  Exploratory measure: brain-derived neurotrophic factor polymorphisms of participants, involved in differential Transcranial direct current stimulation response, will be assess.
Hormonal stress reactivity | One year
  Cortisol level will be measured
Assessment of Cytoplasmic catechol-O-methyltransferase polymorphisms before and after transcranial direct current stimulation. | One year
  Exploratory measure: Cytoplasmic catechol-O-methyltransferase polymorphisms of participants, involved in differential Transcranial direct current stimulation response, will be assess.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme BRUNELIN, PhD, Study Director — Vinatier Hospital PsyR2 Team
Locations (1):
- Ch Le Vinatier, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No